CLINICAL TRIAL: NCT06144671
Title: A Single-Arm Phase I/II Clinical Study of Autologous Tumor-Infiltrating Lymphocyte Injection (GT201) for The Treatment Of Advanced Solid Tumors
Brief Title: GT201 Injection For The Treatment Of Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Grit Biotechnology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GT-CD-CHN-201-01
Record Dates: First submitted 2023-10-20; First posted 2023-11-22 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-10

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GT201 treatment group (Experimental): GT201 5E9（5×10^9）;GT201 1E10（1×10^10）;GT201 5E10（5×10^10）.
  Interventions: Drug: GT201

INTERVENTIONS:
Drug: GT201 — Autologous tumor infiltrating lymphocyte injection

SUMMARY:
Expected to complete 7 to 18 evaluable subjects (patients with advanced solid tumors)，3 dose groups.A modified "3+3" dose-escalation design is utilized,This includes both accelerated dose escalation and traditional "3+3" dose escalation.The first dose group is accelerated titration,The first dose group is an accelerated titration of 1 to 6 evaluable subjects;The second and third dose groups are based on the traditional "3+3" dose-escalation principle,The second and third dose groups are based on the traditional "3+3" dose-escalation principle, with 3 to 6 evaluable subjects enrolled respectively.

ELIGIBILITY:
Inclusion Criteria:

* 1. The Patients (or legally authorized representative) Patients (or legally authorized representative) must have the ability to understand the requirements of the study, have provided written informed consent as evidenced by signature on an informed consent form (ICF) approved by an Institutional Review Board/Independent Ethics Committee (IRB/IEC), must have the ability to understand the requirements of the study;
* 2.Must have a confirmed diagnosis of malignancy of their receptive histologies or cytologies;
* 3.At least one resectable lesion (preferably superficial metastatic lymph nodes) that has not been treated with radiation and has not received other local therapies. The separated tissues ≥1.0cm^3 (either of single lesion origin or multiple lesions combined) for the preparation of autologous tumor-infiltrating lymphocytes. Minimally invasive treatment where possible.

Exclusion Criteria:

* 1.The patient who has any active autoimmune disease, history of autoimmune disease, need for systemic steroid hormones or a condition requiring immunosuppressive drug therapy (>10 mg/day of prednisone or equivalent hormone);
* 2. Arterial/venous thrombotic events within 3 months prior to enrollment, such as: cerebrovascular accident, deep vein thrombosis and pulmonary embolism occurring;
* 3. Patients who have refractory or intractable epilepsy, poorly controlled hydrothorax, hydrops abdominis, pericardial effusion or IL-2 contraindications;
* 4. Participate in other clinical trials within 4 weeks prior to the first dose of this study, or planning to participate in this study and other clinical trials at the same;
* 5. Patients who have received allogeneic bone marrow transplantation or an organ allograft;
* 6.Patients who have a history of hypersensitivity to any component or excipient of study drugs: autologous tumor infiltrating lymphocytes, cyclophosphamide, fludarabine, IL-2, dimethyl sulfoxide (DMSO), human serum albumin (HSA), dextran-40 and antibiotics (beta lactam antibiotics, gentamicin).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2026-09-13 (Estimated); Study Completion 2026-09-13 (Estimated)

PRIMARY OUTCOMES:
Safety Profile Measured By Grade ≥ 3 TREAs | 3 years
  Safety Profile Measured By Grade ≥ 3 TREAs for CTCAE 5.0

SECONDARY OUTCOMES:
Tumor imaging to determine changes in tumor size | 3 years
  Tumor imaging determines the changes in tumor size at baseline and after treatment.Tumor imaging evaluation according to RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - The fifth medical center of the General Hospital of the Chinese people's Liberation Army, Beijing, Beijing Municipality
  - Union Hospital Tongji Medical College Huazhong University Of Science And Technology, Wuhan, Hubei
  - Shandong Cancer Hospital, Jinan, Shandong
  - West China Hospital Sichuan University, Chengdu, Sichuan